CLINICAL TRIAL: NCT04003311
Title: Comprehensive® Primary Micro Stem and Comprehensive® Anatomic Versa-Dial Titanium Humeral Heads in Primary and Revision Total Shoulder Arthroplasty
Brief Title: MDR - Comprehensive Primary/Micro Stem & Versa-Dial Ti Humeral Head
Status: Enrolling by invitation | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: MDRG2017-89MS-46E
Record Dates: First submitted 2019-06-18; First posted 2019-07-01 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Shoulder Pain; Shoulder Injuries; Shoulder Fractures; Shoulder Disease; Shoulder Arthritis
MeSH Terms: conditions — Shoulder Pain; Shoulder Injuries; Shoulder Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Comprehensive Primary Micro Stem: Patients that have been implanted with the Comprehensive Primary Micro Stem to repair shoulder malfunction/disease.
  Interventions: Device: Comprehensive Primary Micro Stem
- Comprehensive Anatomic Versa-Dial Titanium Humeral Heads: Patients that have been implanted with the Comprehensive Anatomic Versa-Dial Titanium Humeral Heads to repair shoulder malfunction/disease.
  Interventions: Device: Comprehensive Anatomic Versa-Dial Titanium Humeral Head

INTERVENTIONS:
Device: Comprehensive Primary Micro Stem — Patients that have been implanted with the Comprehensive Primary Micro Stem to repair shoulder malfunction/disease.
  Groups: Comprehensive Primary Micro Stem
Device: Comprehensive Anatomic Versa-Dial Titanium Humeral Head — Patients that have been implanted with the Comprehensive Anatomic Versa-Dial Titanium Humeral head to repair shoulder malfunction/disease.
  Groups: Comprehensive Anatomic Versa-Dial Titanium Humeral Heads

SUMMARY:
The objective of this retrospective/prospective enrollment and prospective follow-up consecutive series PMCF study is to collect data confirming safety, performance and clinical benefits of the Comprehensive Primary Micro Stem and Comprehensive Anatomic Versa-Dial Titanium Humeral Heads when used for primary and revision total shoulder arthroplasty (implants and instrumentation) at 1,3,5,7 and 10 years*. Comprehensive Primary Micro Stem and Comprehensive Anatomic Versa-Dial Titanium Humeral Heads have been on the market since 2007, but have insufficient data to support 10 years of clinical history. Therefore, a prospective aspect to the study will be utilized in order to collect long-term data.

DETAILED DESCRIPTION:
The objective of this retrospective/prospective enrollment and prospective follow-up consecutive series PMCF study is to collect data confirming safety, performance and clinical benefits of the Comprehensive Primary Micro Stem and Comprehensive Anatomic Versa-Dial Titanium Humeral Heads when used for primary and revision total shoulder arthroplasty (implants and instrumentation) at 1,2,3,5,7 and 10 years*. Comprehensive Primary Micro Stem and Comprehensive Anatomic Versa-Dial Titanium Humeral Heads have been on the market since 2007, but have insufficient data to support 10 years of clinical history. Therefore, a prospective aspect to the study will be utilized in order to collect long-term data.

The primary objective of this study is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications, and adverse events. Relation of the events to either implant or instrumentation should be specified.

The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs).

*The most recent available data will be used. If any of the listed time points are not available, data will be used from last available time point and follow-up will move forward at the closest available time point.

ELIGIBILITY:
Inclusion Criteria:

* Study devices must have been implanted following the surgical technique and IFU for the Comprehensive Micro Stem and/or the Comprehensive Anatomic Versa-Dial Humeral Heads
* Patient must be 18 years of age or older.
* Patient must have undergone a primary or revision shoulder arthroplasty with the Comprehensive Micro Stem and/or the Comprehensive Anatomic Versa-Dial Humeral Heads for a cleared indication. Cleared indications include the following:

  * non-inflammatory degenerative joint disease including osteoarthritis and avascular necrosis,
  * rheumatoid arthritis,
  * revision where other devices or treatments have failed,
  * correction of functional deformity,
  * fractures of the proximal humerus where other methods of treatment are deemed inadequate,
  * difficult clinical management problems including cuff arthroplasty where other treatment methods may not be suitable or may be inadequate.

Exclusion Criteria:

* Absolute contraindications include infection, sepsis, and osteomyelitis.
* Relative contraindications include:

  * Uncooperative patient or patient with neurologic disorders who is incapable or unwilling to follow directions
  * Osteoporosis
  * Metabolic disorders which may impair bone formation
  * Osteomalacia
  * Distant foci of infections which may spread to the implant site
  * Rapid joint destruction, marked bone loss or bone resorption apparent on roentgenogram
* Patient is a prisoner.
* Patient is a current alcohol or drug abuser.
* Patient is known to be pregnant or breastfeeding.
* Patient has a psychiatric illness or cognitive deficit that will not allow for proper informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A consecutive series of subjects implanted with the Comprehensive Primary Micro Stem and/or the Comprehensive Anatomic Versa-Dial Titanium Humeral Heads in primary and/or revision total shoulder arthroplasty according to the approved indications.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Estimated)
Dates: Start 2019-12-13 (Actual); Primary Completion 2028-07-29 (Estimated); Study Completion 2028-07-29 (Estimated)

PRIMARY OUTCOMES:
Device Safety assessed through the frequency and incidence of revisions, complications and Adverse Events | Out to 10 years
  The primary objective of this study is the assessment of safety by analyzing implant survivorship. This will be established by recording the incidence and frequency of revisions, complications, and adverse events. Relation of the events to either implant or instrumentation should be specified.

SECONDARY OUTCOMES:
Device Performance and Benefits evaluated through the Oxford Shoulder Score outcome measure. | Out to 10 years
  The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs), through the use of the Oxford Shoulder Score (OSS). The OSS is a 12 item questionnaire, each with 5 potential answers. Patients rate their symptoms from 1 (minimal symptoms) to 5 (severe symptoms). The combined total gives a minimum score of 12 and a maximum of 60. Higher scores in the OSS imply worse functionality.
Device Performance and Benefits evaluated through the Patient Assessment Questionnaire. | Out to 10 years
  The secondary objective is the assessment of performance and clinical benefits by recording patient-reported clinical outcomes measures (PROMs), through the use of the Patient Assessment Questionnaire where adverse events and/or complications (yes or no), patient's activity level with regard to operative side, based on the UCLA Activity Score(wholly inactive 10, mostly inactive 9, sometimes participates in mild activities 8, regularly participates in mild activities 7, sometimes participates in moderate activities 6, regularly participates in moderate activities 5, regularly participates in active events 4, regularly participates in very active events 3, sometimes participates in impact sports 2, regularly participates in impact sports 1, or not recorded), and the Reported Score if Individual Scores are not available of the Oxford Shoulder Score. The UCLA Activity score rating is from 10 being the best outcome score, and 1 being the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Erin Osborn, Study Director — Zimmer Biomet
Locations (4):
- United States (4):
  - Shoulder Clinic of Idaho, Boise, Idaho
  - Beaumont Health, Royal Oak, Michigan
  - University of Rochester, Rochester, New York
  - Department of Orthopaedics & Rehabilitation The Larner College of Medicine at The University of Vermont, Burlington, Vermont

IPD SHARING:
Plan to Share IPD: No